| Official Title: | Decision Support for Smoking Cessation in Young Adults With |
|---|---|
| | Severe Mental Illness |
| NCT number: | NCT01779440 |
| <b>Document Type:</b> | Study Protocol |
| Date of the | November 24, 2015 |
| Document: | |

## Summary:

Up to 77% of young people with severe mental illnesses smoke [1-4], a rate that is up to <u>five times higher</u> than the rate of daily smoking in other young adults [5, 6]. Contrary to popular belief, smoking tobacco *does not* provide any benefit for mental illness symptom control [7]. People with severe mental illnesses (SMI: schizophrenia and severe mood disorders) are dying, on average, <u>25 years earlier</u> than those without SMI [8, 9]. Much of this early mortality is due to higher rates of heart and lung diseases, cancers, strokes, and diabetes [8-14].

Cessation of smoking in these transition-age young adults can prevent cancer and increase life expectancy to that of non-smokers [15]. Combination treatments are effective in this group [16-21] and therefore key to improving outcomes, but few SMI smokers use them [22-25] despite their interest in quitting [26]. Motivational interventions for cessation increase interest in quitting [24, 27, 28], but <u>public mental health clinicians do not deliver them</u> [23, 29, 30], in part due to economic reasons [31, 32]. Thus cost effective methods to deliver motivational interventions to engage young smokers with SMI into treatment are needed.

To address this gap, we have developed an <u>electronic decision support system</u> (EDSS) for smoking cessation that is specifically tailored for smokers with SMI, who tend to have cognitive deficits and limited computer experience [34]. Similar to

EDSSs developed for other health problems [39], this EDSS provides information and motivational exercises within an easy-to-use, web-based computer program that can be used with minimal or no staff assistance. Initial piloting of the EDSS in <a href="middle-aged">middle-aged</a> SMI smokers showed excellent usability and promising efficacy [33]. <a href="Pilot-testing among young patients suggested that the EDSS increased motivation to quit smoking and provided direction to adapt the format and content of the EDSS for young SMI smokers.

The purpose of this proposal is to further develop the motivational decision support system and to test its ability to motivate <u>young smokers with SMI to quit smoking with cessation treatment</u>.

## The study aims are:

- **Aim 1.** To identify beliefs related to: cessation treatment, social norms for cessation treatment, and perceptions of behavioral control regarding cessation treatment, among young smokers with SMI.
- **Aim 2.** To adapt and complete the development of an EDSS for young smokers with SMI by adding features designed to change salient beliefs identified in Aim 1.
- **Aim 3.** To conduct usability testing of the new EDSS in young smokers with SMI.
- **Aim 4.** To pilot test, using a small randomized, controlled trial, the ability of the new EDSS to change treatment beliefs and to engage young smokers with SMI into cessation treatment. We will also recruit a minimal assessment control group.

## References

- 1. McEvoy, J. and C. Brown, *Smoking in first-episode patients with schizophrenia*. American Journal of Psychiatry, 1999. **156**(7): p. 1120-1121.
- 2. Barnes, T.R.E., et al., *Comorbid substance use and age at onset of schizophrenia*. British Journal of Psychiatry, 2006. **188**: p. 237-42.
- 3. Wade, D., et al., *Course of substance misuse and daily tobacco use in first episode psychosis.* Schizophrenia Research, 2006. **81**: p. 145-50.
- 4. Vanable, P.A., et al., *Smoking among psychiatric outpatients: relationship to substance use, diagnosis, and illness severity.* Psychology of Addictive Behaviors, 2003. **17**(4): p. 259-265.

- 5. Hu, M.-C., M. Davies, and D.B. Kandel, *Epidemiology and correlates of daily smoking and nicotine dependence aong young adults in the United States.* American Journal of Public Health, 2006. **96**: p. 299-308.
- 6. Annonymous, *Cigarette use among high school students --- United States, 1991--2007.* MMWR Morbidity & Mortality Weekly Report, 2008. **57**(25): p. 689-691.
- 7. Hamera, E., J.K. Schneider, and S. Deviney, *Alcohol, cannabis, nicotine, and caffeine use and symptom distress in schizophrenia.* Journal of Nervous and Mental Disease, 1995. **183**: p. 559-565.
- 8. Williams, J.M., et al., *Comparison of two intensities of tobacco dependence counseling in schizophrenia and schizoaffective disorder.* Journal Substance Abuse Treatment, 2010. **38**(4): p. 384-93.
- 9. Colton, C.W. and R.W. Manderscheid, *Congruencies in increased mortality rates, years of potential life lost, and causes of death among public mental health clients in eight states.* Preventing Chronic Disease, 2006. **3**(2): p. 1-14.
- 10. Mauer, B., *Morbidity and mortality in people with serious mental illness*, in *Technical Reports*, J. Parks, et al., Editors. 2006, National Association of State Mental Health Program Directors, Medical Directors Council: Alexandria.
- 11. Carney, C.P., L. Jones, and R.F. Woolson, *Medical comorbidity in women and men with schizophrenia: a population-based controlled study.* J Gen Intern Med, 2006. **21**(11): p. 1133-7.
- 12. Carney, C.P. and L.E. Jones, *Medical comorbidity in women and men with bipolar disorders: a population-based controlled study.* Psychosom Med, 2006. **68**(5): p. 684-91.
- 13. Jones, D.R., et al., *Prevalence, severity, and co-occurrence of chronic physical health problems of persons with serious mental illness.* Psychiatric Services, 2004. **55**(11): p. 1250-7.
- 14. Brown, S., H. Inskip, and B. Barraclough, *Causes of the excess mortality of schizophrenia*. British Journal of Psychiatry., 2000. **177**: p. 212-7.
- 15. Dickey, B., et al., *Medical morbidity, mental illness, and substance use disorders.* Psychiatric Services, 2002. **53**(7): p. 861-867.
- Doll, R., et al., *Mortality in relation to smoking: 50 years' observations on male British doctors.* BMJ, 2004. **26**: p. 1519-28.
- 17. Fiore, M.C., et al., *Treating tobacco use and dependence: 2008 update Clinical practice guideline*. 2008, Rockville, MD: U.S. Department of Health and Human Services. Public Health Service.
- 18. Dixon, L., et al., *Correlates of severity of smoking among persons with severe mental illness.* American Journal on Addictions, 2007. **16**(2): p. 101-10.
- 19. Moeller-Saxone, K., *Cigarette smoking and interest in quitting among consumers at a psychiatric disability rehabilitation and support service in Victoria.* Australian & New Zealand Journal of Public Health., 2008. **32**(5): p. 479-481.
- 20. Siru, R., G.K. Hulse, and R.J. Tait, *Assessing motivation to quit smoking in people with mental illness: a review.* Addiction, 2009. **104**(5): p. 719-33.
- 21. Etter, M., et al., *Stages of change in smokers with schizophrenia or schizoaffective disorder and in the general population.* Schizophrenia Bulletin, 2004. **30**(2): p. 459-68.
- 22. Gershon Grand, R.B., et al., *Short-term naturalistic treatment outcomes in cigarette smokers with substance abuse and/or mental illness.* Journal of Clinical Psychiatry, 2007. **68**(6): p. 892-8.
- 23. Ferron, J.C., et al., *A review of research on smoking cessation interventions for adults with schizophrenia spectrum disorders.* Mental Health and Substance Abuse: Dual Diagnosis, 2009. **2**(1): p. 64-79.

- 24. Evins, A.E., et al., A double-blind placebo-controlled trial of bupropion sustained-release for smoking cessation in schizophrenia.[see comment]. Journal of Clinical Psychopharmacology, 2005. **25**(3): p. 218-25.
- 25. George, T.P., et al., *A placebo controlled trial of bupropion for smoking cessation in schizophrenia.* Biological Psychiatry, 2002. **52**: p. 53-61.
- 26. Evins, A.E., et al., *A 12-week double-blind, placebo-controlled study of bupropion sr added to high-dose dual nicotine replacement therapy for smoking cessation or reduction in schizophrenia.* Journal of Clinical Psychopharmacology, 2007. **27**(4): p. 380-6.
- 27. Evins, A.E., et al., *A controlled trial of bupropion added to nicotine patch and behavioral therapy for smoking cessation in adults with unipolar depressive disorders.* Journal of Clinical Psychopharmacology, 2008. **28**(6): p. 660-6.
- 28. Baker, A., et al., *A randomized controlled trial of a smoking cessation intervention among people with a psychotic disorder.* American Journal of Psychiatry, 2006. **163**(11): p. 1934-42.
- 29. Stuyt, E.B., B. Order-Connors, and D.M. Ziedonis, *Addressing tobacco through program and system change in mental health and addiction settings.* Psychiatric Annals, 2003. **33**: p. 446-56.
- 30. Annonymous, *Helping psychiatric patients to stop smoking.* Harvard Mental health letter, 2008. **September**: p. 4-5.
- 31. Schroeder, S.A., *A 51-year-old woman with bipolar disorder who wants to quit smoking.* Journal of the American Medical Association, 2009. **301**(5): p. 522-31.
- 32. Addington, J., et al., *Readiness to stop smoking in schizophrenia*. Canadian Journal of Psychiatry, 1997. **42**: p. 49-52.
- 33. Baker, A., et al., *Characteristics of smokers with a psychotic disorder and implications for smoking interventions.* Psychiatry Research, 2007. **150**(2): p. 141-52.
- 34. Esterberg, M. and M. Compton, *Smoking behavior in persons with schizophrenia-spectrum disorder: a qualitative investigation of the transtheoretical model.* Social Science and Medicine, 2005. **61**(293-303).
- 35. Lucksted, A., L.B. Dixon, and J.B. Sembly, *A focus group pilot study of tobacco smoking among psychosocial rehabilitation clients.* Psychiatric Services, 2000. **51**(12): p. 1544-8.
- 36. Morris, C.D., et al., *What do persons with mental illnesses need to quit smoking? Mental health consumer and provider perspectives.* Psychiatric Rehabilitation Journal, 2009. **32**(4): p. 276-84.
- 37. Davis, K.L., et al., *A qualitative study of smoking maintenance and cessation in persons with serious mental illness.* Journal of Mental Health and Substance Use: Dual Diagnosis, 2010. **3**(2): p. 110-123.
- 38. Tucker, J.S., et al., *Predictors of attempted quitting and cessation among young adult smokers.* Preventive Medicine, 2005. **41**(2): p. 554-61.
- 39. Pirie, P.l., D.M. Murray, and R.V. Luepker, *Gender differences in cigarette smoking and quitting in a cohort of young adults.* 1991(0090-0036 (Print)).
- 40. Agrawal, A., et al., *Correlates of smoking cessation in a nationally representative sample of U.S. adults.* Addict Behay, 2008. **33**(9): p. 1223-6.
- 41. Chen, K. and D.B. Kandel, *The natural history of drug use from adolescence to the mid-thirties in a general population sample.* Am J Public Health, 1995. **85**(1): p. 41-7.
- 42. Vangeli, E. and R. West, *Sociodemographic differences in triggers to quit smoking: findings from a national survey.* Tobacco Control, 2008. **17**(6): p. 410-15.
- 43. Gilpin, E., et al., *Reasons smokers give for stopping smoking: do they related to success in stopping?* Tobacco Control, 1992. **1**: p. 256-63.
- 44. Solberg, L.I., et al., *Young adult smokers: are they different?* American Journal of Managed Care, 2007. **13**(11): p. 626-32.

- 45. DeBernardo, R.L., et al., *An E-mail assessment of undergraduates' attitudes toward smoking.* Journal of American College Health, 1999. **48**(2): p. 61-6.
- 46. Hines, D., Young smokers' attitudes about methods for quitting smoking: Barriers and benefits to using assisted methods. Addictive Behaviors. **21**(4): p. 531-535.
- 47. Millstein, S.G. and B.L. Halpern-Felsher, *Judgements about risk and perceived invulnerability in adolescents and young adults.* Journal of Research on Adolescence, 2002. **12**(4): p. 399-422.
- 48. Davis, M., *Addressing the needs of youth in transition to adulthood.* Administration & Policy in Mental Health, 2003. **30**(6): p. 495-509.
- 49. Webb, T.L., et al., *Using the internet to promote health behavior change: a systematic review and meta-analysis of the impact of theoretical basis, use of behavior change techniques, and mode of delivery on efficacy.* Journal of Medical Internet Research, 2010. **12**(1): p. e4.
- 50. Ajzen, I., *The theory of planned behavior*. Organizational Behavior and Human Decision Processes, 1991. **50**: p. 179-211.
- 51. Godin, G. and K. Gerjo, *The Theory of Planned Behavior: A review of its appications to health-related behaviors.* American Journal of Health Promotion, 1996. **11**(2): p. 87-98.
- 52. Norman, P., M. Conner, and R. Bell, *The Theory of Planned Behavior and smoking cessation.* Health Psychology, 1999. **18**(1): p. 89-94.
- 53. Boissonneault, E. and G. Godin, *The prediction of intention to smoke only in designated work site areas.* Journal of Occupational Medicine, 1990. **32**: p. 621-4.
- 54. Borland, R., et al., *Predicting attempts and sustained cessation of smoking after the introduction of workplace smoking bans.* Health Psychology, 1991. **10**: p. 336-42.
- 55. De Vries, H., M. Kijkstra, and P. Kuhlman, *Self-efficacy: the third factor besides attitude and subjective norm as predictor of behavioral intentions.* Health Education Research, 1988. **3**: p. 273-82.
- 56. Godin, G. and L. Lepage, *Understanding the intentions of pregnant nullipara to not smoke cigarettes after childbirth.* Journal of Drug Education, 1988. **18**: p. 115-24.
- 57. Godin, G., et al., *Predictors of smoking behavior: an application of Ajzen's theroy of planned behavior.* British Journal of Addiction, 1992. **87**: p. 1335-1343.
- 58. Steinberg, M.L., et al., *Motivational interviewing with personalized feedback: a brief intervention for motivating smokers with schizophrenia to seek treatment for tobacco dependence.* Journal of Consulting and Clinical Psychology, 2004. **72**(4): p. 723-8.
- 59. Cather, C., et al. A randomized controlled trial of motivational interviewing compared to psychoeducation for smoking pre-contemplators with severe mental illness. in Society for Research on Nicotine and Tobacco. 2010. Baltimore.
- 60. Williams, J.M., et al., *A wellness approach to addressing tobacco in mental health settings: learning aobut healthy living.* American Journal of Psychiaric Rehabilitation, 2009. **12**: p. 352-369.
- 61. Levit, K.R., et al., *Future funding for mental health and substance abuse: increasing burdens for the public sector.* Health Aff (Millwood), 2008. **27**(6): p. w513-22.
- 62. Truffer, C.J., et al., *Health spending projections through 2019: the recession's impact continues.* Health Aff (Millwood). **29**(3): p. 522-9.
- 63. Brunette, M.F., et al., *Implementation of Integrated Dual Disorder Treatment:*
- *A Qualitative Analysis of Facilitators and Barriers.* Psychiatric Services, 2008. **59**: p. 989-95.
- 64. Weinberger, A.H., et al., *Survey of clinician attitudes toward smoking cessation for psychiatric and substance abusing clients.* Journal of Addictive Diseases, 2008. **27**(1): p. 55.
- 65. Stead, L.F., R. Perera, and T. Lancaster, *Telephone counseling for smoking cessation (review)*. Cochrane Database of Systematic Reviews, 2006. **3**.
- 66. Lichtenstein, E., S.H. Zhu, and G.J. Tedeschi, *Smoking cessation Quitlines: An underrecognized intervention success story.* American Psychologist, 2010. **65**: p. 252-61.

- 67. Green, M.J., et al., Effect of a Computer-Based Decision Aid on Knowledge, Perceptions, and Intentions About Genetic Testing for Breast Cancer Susceptibility: A Randomized Controlled Trial. Journal of American Medical Association, 2004. **292**(4): p. 442-452.
- 68. Valimaki, M., et al., *Design and development process of patient-centered computer-based support system for patients with schizophrenia spectrum psychosis.* Inform Health Soc Care, 2008. **33**(2): p. 113-23.
- 69. Myung, S.K., et al., *Effects of Web- and computer-based smoking cessation programs: meta-analysis of randomized controlled trials.* Arch Intern Med, 2009. **169**(10): p. 929-37.
- 70. Annonymous, *Research-based web design & usability guidelines*, Washington, D.C.: United States Department of Health and Human Services.
- 71. Ueland, T. and B.R. Rund, *Cognitive remediation for adolescents with early onset psychosis: a 1-year follow-up study.* Acta Psychiatrica Scandinavica, 2005. **111**: p. 193-201.
- 72. Wolford, G.L., et al., *Evaluation of methods for detecting substance use disorder in persons with severe mental illness.* Psychology of Addictive Behaviors, 1999. **13**: p. 313-326.
- 73. Rotondi, A.J., et al., *Designing websites for persons with cognitive deficits: Design and usability of a psychoeducational interevention for person with severe mental illness.* Psychological Services, 2007. **4**(3): p. 202-24.
- 74. Andrews, S., et al., *Developing web-based online support tools: The Dartmouth decision support softward.* Psychiatric Rehabilitation Journal, In press.
- 75. Drake, R.E., et al., *The Thresholds-Dartmouth partnership and research on shared decision making.* Psychiatric Services, 2009. **60**(2): p. 142-4.
- 76. O'Connor, A.M., et al., *Decision aids for people facing health treatment or screening decisions.* Cochrane Database of Systematic Reviews, 2009(3): p. CD001431.
- 77. Brunette, M.F., et al., *Testing an electronic decision support system to increase motivation for smoking cessation among persons with severe mental illness.* Psychiatric Services, In press.
- 78. Ferron, J.C. and M.F. Brunette, *The development and usability testing of website to educate and engage people with severe mental illness into smoking cessation treatment.* Psychiatric Rehabilitation Journal, Submitted.
- 79. Barbour, R.S. and M. Barbour, *Evaluating and synthesizing qualitative research: The need to develop a distinctive approach.* Journal of Evaluation in Clinical Practice, 2003. **9**: p. 179-186.
- 80. Miles, M. and A. Huberman, *Qualitative data analysis*. 1994, Thousand Oaks California: Sage.
- 81. Ferron, J.C., et al., *Longitudinal course of smoking and quit attempts in clients with co-occurring Severe mental illness and substance use disorders.* Psychiatric Services, Submitted.
- 82. Miller, W.R. and S. Rollnick, eds. *Motivational Interviewing: Preparing People for Change.* Second ed. 2002, Guilford Press: New York.
- 83. O'Connor, A. and M.J. Jacobsen. *Workbook on developing and evaluating patient decision aids.* 2003 [cited.
- 84. Javors, M.A., J.P. Hatch, and R.J. Lamb, *Cut-off levels for breath carbon monoxide as a marker for cigarette smoking.* Addiction, 2005. **100**(2): p. 159-67.
- 85. Ziedonis, D.M. and K. Trudeau, *Motivation to quit using substances among individuals with schizophrenia: Implications for a motivation-based treatment model.* Schizophrenia Bulletin, 1997. **23**: p. 229-238.
- 86. Ericsson, K.A. and H.A. Simon, *Protocol analysis: verbal reports as data.* 1993, Cambridge, MA: MIT Press.
- 87. Rubin, J. and D. Chisnell, *Handbook of Usability Testing, 2nd Edition*. Wiley technical communication library. 2008: Wiley.
- 88. Ajzen, I. *Behavioral interventions based on the theory of planned behavior*. 2006 [cited; Available from: http://www.people.umass.edu/aizen/pdf/tpb.intervention.pdf.
- 89. Francis, J.J., et al., *Constructing questionnaires based on the Theory of Planned Behavior*. 2004, Newcastle Upon Tyne, U.K.: Center for Health Services Research.

- 90. Ajzen, I. *Constructing a TpB Questionnaire: Conceptual and methodological considerations.* 2006 2006 [cited 2010 May 2, 2010].
- 91. Durkin, S.J., L. Biener, and M.A. Wakefield, *Effects of different types of antismoking as on reducing disparities in smoking cessation among socioeconomic groups.* American Journal of Public Health, 2009. **99**(12): p. 2217-2223.
- 92. Edwards, A., G. Elwyn, and A. Mulley, *Explaining risks: turning numberical data into meaningful pictures*. BMJ, 2002. **324**: p. 827-830.
- 93. Tversky, A. and D. Kahneman, *The framing of decisions and the psychology of choice.* Science, 1981. **211**: p. 453-58.
- 94. Rothman, A.J. and P. Salovey, *Shaping perceptions to motivate health behavior: The role of message framing.* Psychological Bulletin, 1997. **121**(1): p. 3-19.
- 95. Simonsen, E., et al., *Clinical epidemiological first-episode psychosis: 1- year outcome and predictors.* Acta Psychiatrica Scandinavia, 2007. **116**(1): p. 54-61.
- 96. Wilson, D.K., K.A. Wallston, and J.E. King, *Effects of contract framing, motivation to quit and self-efficacy on smoking reduction.* Journal of Applied Social Psychology, 2006. **20**(7): p. 531-547.
- 97. Toll, B.A., et al., *Comparing gain- and loss-framed messages for smoking cessation with sustained-release bupropion: A randomized controlled trial.* Psychology of Addictive Behaviors, 2007. **21**(4): p. 534-544.
- 98. Edwards, A., et al., *Presenting risk information to people with diabetes: evaluating effects and preferences for different formats by a web-based randomised controlled trial.* Patient Education & Counseling, 2006. **63**(3): p. 336-49.
- 99. Edwards, A. and G. Elwyn, *Understanding risk and lessons for clinical risk communication about treatment preferences.* Quality in Health Care, 2001. **10(Suppl 1)**: p. i9-i13.
- 100. Gough, B., et al., *Why do young adult smokers continue to smoke despite the health risks? A focus group study.* Psychology & Health, 2009. **24**(2): p. 203-20.
- 101. Klein, W.M., L.E. Zajac, and M.M. Monin, *Worry as a moderator of the association between risk perceptions and quitting intentions in young adult and adult smokers.* Annals of Behavioral Medicine, 2009. **38**(3): p. 256-61.
- 102. Etcheverry, P.E. and C.R. Agnew, Romantic partner and friend influences on young adult cigarette smoking: comparing close others' smoking and injunctive norms over time. Psychology Addictive Behaviors, 2008. **22**(3): p. 313-25.
- 103. Green, K.J., et al., *Peer and role model influences for cigarette smoking in a young adult military population.* Nicotine & Tobacco Research, 2008. **10**(10): p. 1533-41.
- Hammond, D., et al., *Tobacco denormalization and industry beliefs among smokers from four countries.* American Journal of Preventive Medicine, 2006. **31**(3): p. 225-232.
- 105. Ling, P.M., T.B. Neilands, and S.A. Glantz, *Young adult smoking behavior: a national survey.* American Journal of Preventive Medicine, 2009. **36**(5): p. 389-394 e2.
- 106. Sussman, S., et al., *Attitudes of adolescents towards smoking cessation.* Preventive Medicine, 1998. **27**: p. A19-A28.
- 107. Stoddard, J.L., E.M. Augustson, and P.L. Mabry, *The importance of usability testing in the development of an internet-based smoking cessation treatment resource.* Nicotine Tob Res, 2006. **8 Suppl 1**: p. S87-93.
- 108. Evans, R., et al., *Toward a model for field-testing patient decision-support technologies: a qualitative field-testing study.* Journal of Medical Internet Research, 2007. **9**(3): p. e21.
- 109. van Someren, M.W., Y.F. Barnard, and J.A.C. Sandberg, *The think aloud method A practical guide to modelling cognitive processes*. 1994, London: Academic Press.
- 110. Davis, F.D., *Perceived usefulness, perceived ease of use, and user acceptance and information technology.* MIS Quarterly, 1989. **13**(3): p. 319-340.

- 111. Tohen, M., et al., *The McLean-Harvard First-episode project: 6-month symptomsatic and fucntional outcome in affective and nonaffective psychosis.* Biological Psychiatry, 2000. **48**: p. 467-476.
- 112. Hasin, D., et al., *Epidemiology of major depressive disorder Results from the National Epidemionlogic Survey on Alcoholism and Related Conditions.* Archives General Psychiatry, 2005. **62**: p. 1097-1106.
- 113. Bertelsen, M., et al., *Five-year follow-up of a randomized multicenter trial of intensive early intervention vs standard treatment for patients with a first episode of psychotic illness: the OPUS trial.* Arch Gen Psychiatry, 2008. **65**(7): p. 762-71.
- 114. Shern, D.L., N.Z. Wilson, and A.S. Coen, *Client outcomes II: Longitudinal client data from the Colorado treatment outcome study.* Milbank Quarterly, 1994. **72**(1): p. 123-148.
- 115. Conrad, K.J., et al., *Reliability and validity of a modified Coloarado symptom index in a national homeless sample.* Mental Health Services Research, 2001. **3**(3): p. 141-53.
- 116. Agosti, V. and F.R. Levin, *Does remission from alcohol and drug use disorders increase the likelihood of smoking cessation among nicotine dependent young adults?* Social Psychiatry and Psychiatric Epidemiology, 2009. **44**: p. 120-124.
- 117. Stapleton, J.A., F. Keaney, and G. Sutherland, *Illicit drug use as a predictor of smoking cessation treatment outcome*. Nicotine & Tobacco Research, 2009. **11**(2): p. 685-89.
- 118. Prochaska, J.J., K. Delucchi, and S.M. Hall, *A meta-analysis of smoking cessation interventions with individuals in substance abuse treatment or recovery.* J Consult Clin Psychol, 2004. **72**(6): p. 1144-56.
- 119. Baca, C.T. and C.E. Yahne, *Smoking cessation during substance abuse treatment: what you need to know.* Journal of Substance Abuse Treatment, 2009. **36**(2): p. 205-19.
- 120. Hall, S.M. and J.J. Prochaska, *Treatment of smokers with co-occurring disorders: emphasis on integration in mental health and addiction treatment settings.* Annual Review of Clinical Psychology, 2009. **5**: p. 409-31.
- 121. Einarson, A. and S. Riordan, *Smoking in pregnancy and lactation: a review of risks and cessation strategies.* European Journal of Clinical Pharmacology, 2009. **65**(4): p. 325-30.
- Lumley, J., et al., *Interventions for promoting smoking cessation during pregnancy.* Cochrane Database of Systematic Reviews, 2009(3): p. CD001055.
- 123. Keefe, R.S., et al., *The Brief Assessment of Cognition in Schizophrenia: reliability, sensitively and comparison with a standard neurocognitive battery.* Schizophrenia Research, 2004. **68**(2-3): p. 283-97.
- Williams, J.M. and D. Ziedonis, *Addressing tobacco among individuals with a mental illness or an addiction.* Addict Behav, 2004. **29**(6): p. 1067-83.
- 125. Williams, J.M. and J. Foulds, *Successful tobacco dependence treatment in schizophrenia*. Am J Psychiatry, 2007. **164**(2): p. 222-7; quiz 373.
- 126. Gelenberg, A.J., et al., *Smoking cessation in patients with psychiatric disorders.* Journal of Clinical Psychiatry, 2007. **68**(9): p. 1404-10.
- 127. Cather, C., V.K. Mays, and J.D. Gottlieb, *13-week cognitive behavioal therpay group treatment for smokin gcessation designed to be used with individuals wiht schizophrenia paritcipating in the varenicline study.* 2007.
- 128. Culhane, M.A., et al., *Predictors of early abstinence in smokers with schizophrenia.* Journal of Clinical Psychiatry, 2008. **69**(11): p. 1743-50.
- 129. Brown, R.A., et al., *Reliability and Validity of Smoking Timeline Follow-Back Interview.* Psychology of Addictive Behaviors, 1998. **12**(2): p. 101-112.
- 130. Sobell, L.C. and M.B. Sobell, *Alcohol Timeline Followback (TLFB) Users' Manual.* 1996, Toronto, Canada: Addiction Research Foundation.
- 131. Carey, K., K. Cocco, and J. Simons, *Concurrent validity of clinicians' ratings of substance abuse among psychiatric outpatients.* Psychiatric Services, 1996. **47**: p. 842-847.

- 132. Jarvis, M.J., M.A. Russell, and Y. Saloojee, *Expired air carbon monoxide: a simple breath test of tobacco smoke intake.* Br Med J, 1980. **281**(6238): p. 484-5.
- 133. Benowitz, N.L., et al., *Biochemical verification of tobacco use and cessation.* Nicotine & Tobacco Research, 2002. **4**.
- 134. Fagerström, K.O., Measuring degree of physical dependency to tobacco smoking with reference to individualization of treatment. Addictive Behaviors, 1978. 3: p. 235-241.
- 135. Weinberger, A.H., et al., *Reliability of the Fagerstrom Test for Nicotine Dependence, Minnesota Nicotine Withdrawal Scale, and Tiffany Questionnaire for Smoking Urges in smokers with and without schizophrenia.* Drug and Alcohol Dependence, 2007. **86**: p. 278-82.
- 136. Sobell, L.C., et al., *Comparison of a quick drinking screen with timeline followback for individuals with alcohol problems.* Journal of Studies on Alcohol, 2003. **64**: p. 858-861.
- 137. Hosmer, D.W. and S. Lemneshow, *Applied Logistic Regression*. 1989, New York: J. Wiley & Sons.
- 138. Brunette MF, Ferron JC, Drake RE, Devitt TS, Geiger PT, McHugo GJ, et al. Carbon monoxide feedback in a motivational decision support system for nicotine dependence among smokers with severe mental illnesses. Journal of substance abuse treatment. 2013;45(4):319-24. Epub 2013/05/28. doi: 10.1016/j.jsat.2013.04.005. PubMed PMID: 23706623.
- 139. Ferron JC, Brunette MF, McGurk S, H. X, Frounfelker R, Cook JA. Do symptoms and cognitive problems affect the use and efficacy of a web-based decision support system for smokers with serious mental illness? Journal of Dual Diagnosis. 2012;8(4):315-25.
- 140. Graham, A.W., *Screening for alcoholism by life-style risk assessment in a community hospital.* Archives of Internal Medicine, 1991. **151**: p. 958-964.